CLINICAL TRIAL: NCT04262427
Title: The CAPER Study: A Phase Ib Clinical Trial of Cyclophosphamide And PEmbrolizumab in Metastatic Renal Cell Carcinoma (RCC) (CAPER Trial)
Brief Title: The CAPER Trial: A Phase Ib Clinical Trial of Cyclophosphamide And PEmbrolizumab in Metastatic Renal Cell Carcinoma
Acronym: CAPER
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); University of Liverpool (Other); University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFTSp148; 2018-004314-17 (EudraCT Number)
Record Dates: First submitted 2020-01-28; First posted 2020-02-10 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Cyclophosphamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group Assignment (Experimental): Cyclophosphamide 50mg PO OD for 3 weeks as monotherapy followed by cyclophosphamide 50mg PO OD with pembrolizumab 200mg IV every 3 weeks
  Interventions: Drug: Cyclophosphamide 50mg; Drug: Pembrolizumab 25 mg/1 ML Intravenous Solution [KEYTRUDA]

INTERVENTIONS:
Drug: Cyclophosphamide 50mg — cytotoxic chemotherapy
  Other Names: cyclophosphamide monohydrate
Drug: Pembrolizumab 25 mg/1 ML Intravenous Solution [KEYTRUDA] — potent humanized immunoglobulin (Ig) G4 monoclonal antibody (mAb) with high specificity of binding to the programmed cell death 1 (PD-1) receptor
  Other Names: Keytruda, MK-3475

SUMMARY:
This is an open label investigator initiated Phase Ib study of combination pembrolizumab (Keytruda), 200mg IV 3 weekly (Q3W) with 50mg oral cyclophosphamide daily (OD) in metastatic renal cell carcinoma patients. 21 patients will be recruited within the United Kingdom (UK) will to examine the efficacy of the combination for up to 35 administrations (2 years). This study will be conducted in compliance with Good Clinical Practice (GCP) and all relevant regulations.

DETAILED DESCRIPTION:
The CAPER Trial will be looking at patients with locally advanced (inoperable) or metastatic clear cell renal cell carcinoma who have had previous treatment with immunotherapy and have experienced disease progression. Immunotherapies aim to boost the body's natural defences to fight cancer, however the tumour micro-environment may significantly impact how effective this approach will be at reducing cancer growth and spread. The CAPER trial aims to evaluate whether oral metronomic cyclophosphamide (50mg once daily) can alter the tumour environment and ultimately lead to responses to pembrolizumab in patients who have failed prior immunotherapy.

Patients who join the study will initially take cyclophosphamide 50mg tablets once a day for 21 days during the 'run-in period'. Following this, they will continue with cyclophosphamide 50mg daily alongside intravenous pembrolizumab treatment administered once every 3 weeks. Patients will continue both treatments until the occurrence of either disease progression, unexpected toxicity, patient withdrawal, or completion of 24 months of treatment.

Patients will undergo CT scanning to evaluate response every 9 weeks during trial treatment.

Research biopsies will be taken at baseline (prior to treatment), after the 21 day run-in period on oral cyclophosphamide, and at the time of the first CT scan (week 9 on treatment). Patients will also have additional research blood samples collected at serial timepoints whilst on treatment. The biopsy and blood samples will allow evaluation of the changes induced by cyclophosphamide and pembrolizumab within the tumour microenvironment as well as changes in circulating factors such as cytokines.

ELIGIBILITY:
INCLUSION CRITERIA

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Histological confirmation of RCC of predominantly (>50%) clear cell type.
2. Presence of metastatic / locally advanced inoperable disease.
3. Current evidence of disease progression on immuno-oncology (IO) therapy as determined by CT / MRI imaging performed within 28 days prior to the first dose of study drug. Last dose of IO therapy must have been administered within 42 days prior to the first dose of study drug. IO therapy may consist of either:

   1. First-line Ipilimumab / Nivolumab combination OR
   2. Second / Third-line single agent Nivolumab OR
   3. Other PD-1 / PD-L1 / anti-CTLA-4 therapy within a clinical trial
4. Measurable disease according to RECIST version 1.1 criteria.
5. Site(s) of disease which are easily accessible and suitable for repeated biopsies (bone metastases are not suitable as a biopsy site).
6. Provision of archival tumour tissue sample (formalin-fixed paraffin embedded (FFPE) tissue blocks) and a newly obtained core or excisional biopsy of a tumour lesion not previously irradiated.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study drug.
8. Age > 18 years.
9. Have adequate organ function as defined below. Specimens must be collected within 14 days prior to the start of study treatment.

   1. Absolute neutrophil count (ANC) ≥1.5 x109/L
   2. Platelets ≥100 x109/L
   3. Haemoglobin ≥9.0 g/dL or ≥5.6 mmol/L
   4. Creatinine ≤1.5 × Upper Limit of Normal (ULN) OR Measured or calculated creatinine clearance (CrCl) ≥30 mL/min for participant with creatinine levels OR (Glomerular Filtration Rate (GFR) can also be used in place of creatinine or CrCl >1.5 × institutional ULN
   5. Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
   6. Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
   7. International normalised ratio (INR) OR prothrombin time (PT) / Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
10. Able to take oral medications.
11. Life expectancy of > 6 months in the opinion of the investigator.
12. Male participants must agree to use a form of contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.
13. Female participants are eligible to participate if they are not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
    2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 180 days after the last dose of study treatment.
14. The participant provides written informed consent for the trial including consent to all samples.

EXCLUSION CRITERIA

Participants are excluded from the study if any of the following criteria apply:

1. Treatment with more than one prior line of IO therapy (including previous standard of care and trial treatments).
2. High burden / symptomatic disease which in the opinion of the treating investigator requires Tyrosine Kinase Inhibitors (TKI) / alternative therapeutic approach.
3. Prior treatment with either pembrolizumab or cyclophosphamide.
4. Known severe hypersensitivity (≥Grade 3) to pembrolizumab, cyclophosphamide and/or any of their excipients.
5. Prior intolerance to IO therapy (any > Grade 2 toxicity which required permanent IO treatment discontinuation).
6. Ongoing Adverse Events (AEs) due to previous therapies or surgery which have not resolved to ≤ Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy may be eligible.
7. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. levothyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
8. Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisolone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
9. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial transitional cell carcinoma of the bladder / urothelial tract, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
10. Prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS (Central Nervous System) disease.
11. Live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist®) are live attenuated vaccines and are not allowed.
12. Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
13. Known previous or current Central Nervous System (CNS) metastases and/or carcinomatous meningitis. Note: no testing is required.
14. History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
15. Active infection requiring systemic therapy or has had requirement for antibiotics within 14 days prior to first dose of study treatment.
16. Known history of Human Immunodeficiency Virus (HIV). Note: no testing for HIV is required.
17. Known history of Hepatitis B (defined as Hepatitis B surface antigen (HBsAg) reactive) or known active Hepatitis C virus (defined as HCV RNA positive) infection. Note: no testing for Hepatitis B and Hepatitis C is required.
18. Known history of active tuberculosis (Bacillus Tuberculosis, TB). Note: no testing for TB is required.
19. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
20. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
21. Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of trial treatment. Note: WOCBP must have a negative urine pregnancy test within 72 hours prior to trial entry (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2023-10-28 (Estimated); Study Completion 2024-04-28 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From baseline up to 2 years, first documented progression or death
  Occurrence of complete response or partial response as defined by RECIST v1.1 at any point in follow-up until end of study or death. Best Objective Response is the highest value achieved for each patient and will be used for the primary outcome analysis.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the time of first treatment up to 2 years, the time of first documented progression, the censor date in months or death
  To evaluate the median PFS in patients receiving cyclophosphamide and pembrolizumab in combination. PFS events are defined as either disease progression or death from any cause. The event date used for analysis will be the first occurrence of either disease progression or death and the analysis will use the following formula:
  Progression-free survival (months) = (exit date - date of first treatment)/30.4
Overall Survival (OS) | From first treatment up to 2 years or death by any cause in months
  To evaluate the median OS in patients receiving cyclophosphamide and pembrolizumab in combination. OS events are defined as death from any cause. The event date used for analysis will be the confirmed date of death and the analysis will use the following formula:
  Overall Survival (months) = (Exit date - date of first treatment)/30.4
Incidence of treatment-emergent adverse events as assessed by occurrence of serious adverse events and adverse events of grade 3 severity and above | From commencement of treatment to 30 days post cessation of treatment
  To evaluate the safety profile of the combination of oral cyclophosphamide and pembrolizumab. The number of patients reporting Serious Adverse Events (SAEs) and Grade 3 or higher toxicity will be summarised overall and by preferred term (if severity is missing, the worst case will be assumed).

CONTACTS AND LOCATIONS:
Overall Officials: Tom Waddell, Principal Investigator — The Christie NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Western General Hospital, NHS Lothian, Edinburgh
  - Royal Marsden Hospital NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Undecided